CLINICAL TRIAL: NCT02072694
Title: Cerebral Perfusion Changes in Obese Subjects After Administration of 75 Grams of Glucose. A SPECT, Controlled, Blinded and Randomized Study.
Brief Title: Cerebral Blood Flow Changes in People With Obesity After Glucose Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Julio Sergio Marchini, Full Professor of Internal Medicine Department at Ribeirão Preto Medical School, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Process HCRP: 12241/2010; CAAE - 0426.0.004.000-10 (Registry Identifier: Sistema Nacional de Informações sobre Ética em Pesquisa)
Record Dates: First submitted 2014-02-22; First posted 2014-02-26 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: Obesity; Single Photon Emission Computed Tomography; Functional Neuroimaging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 75 grams of glucose plus water solution (Experimental): In the group with 10 volunteers with obesity, some of them are submitted first to the 75 grams of glucose plus water solution (meal challenge) and in another time to only water.
  Also, in the group with 10 volunteers without obesity, some of them are submitted first to the 75 grams of glucose plus water solution (meal challenge) and in another time to only water.
  Interventions: Other: 75 grams of glucose plus water solution; Other: Pure water
- Pure water. (Placebo Comparator): In the same group with 10 volunteers with obesity, some of them are submitted first to only water (control) and in another time to the 75 grams of glucose plus water solution (meal challenge).
  Also, in the same group with 10 volunteers without obesity, some of them are submitted first to only water (control) and in another time to the 75 grams of glucose plus water solution (meal challenge).
  Interventions: Other: 75 grams of glucose plus water solution; Other: Pure water

INTERVENTIONS:
Other: 75 grams of glucose plus water solution — A solution composed by 75 grams of glucose and water at ambient temperature is administered to each volunteer, being of the with obesity group or the without obesity group, as follow:
  * 300 mL final volume of the solution.
  * Time of oral ingestion inferior than 2 minutes.
  * 30 minutes before the radiopharmaceutical injection.
  * 12 hours fasting minimum.
Other: Pure water — Pure water at ambient temperature is administered to each volunteer, being of the with obesity group or the without obesity group, as follow:
  * 300 mL final volume of the solution.
  * Time of oral ingestion inferior than 2 minutes.
  * 30 minutes before the radiopharmaceutical injection.
  * 12 hours fasting minimum.

SUMMARY:
This study evaluates the hypothesis that a meal constituted of only glucose produces differences in the brain blood flow in people with obesity that are not observed in people without obesity. These changes, at least in part, could explain the mechanisms involved in maintenance or development of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Live in Ribeirão Preto, São Paulo - Brazil.
* Age between 18 and 40 years old.
* Female gender.
* Regular menses.
* Weight inferior than 120 Kg and body mass index (BMI) between 30 and 40 kg/m2, for the group with obesity.
* BMI between 18,5 and 24,9 kg/m2, for the group without obesity.

Exclusion Criteria:

* High blood pressure, diabetes, glucose intolerance or impaired fasting glycemia, metabolic syndrome, hypothyroidism and any kidney, liver, heart or neurologic disease.
* Psychiatric disorders, alcoholism, smoking or illicit drug abuse.
* Pregnancy or desire to be pregnant
* Use of medications, excluding contraceptives.
* Contraindication for magnetic resonance imaging.
* Be in treatment for obesity.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Regional cerebral blood flow (rCBF) changes after a meal challenge, measured by Single Single-photon emission computed tomography (SPECT) and statistical parametric mapping. | 30 minutes after a meal challenge (time of radiopharmaceutical injection)
  Using 99m technetium ecd radiopharmaceutical, this study aims to detect rCBF differences between SPECT images performed after a meal challenge composed by 75 grams of glucose and water and also after a challenge constituted by only water (control), both ingested orally. This approach is performed in a group of 10 people with obesity and also in 10 people without obesity.

SECONDARY OUTCOMES:
Blood levels mean differences within both groups, with and without obesity and across these groups, of hormones and metabolites by multiplexed assay using luminex technology and spectrophotometry, respectively. | 30 minutes before, at the time and 30, 60 and 90 minutes after the radiopharmaceutical injection.
  This study looks for mean differences of blood levels within and across groups with and without obesity. The metabolites and hormones/cytokines measured are, respectively: glucose (measured by spectrophotometry), insulin, leptin, amylin, interleukin 6 (IL-6), tumor necrosis factor alpha, active ghrelin, peptide yy (PYY) and pancreatic polypeptide (PP) (multiplexed assay using luminex).
Resting energy expenditure (REE) and body composition measurements by indirect calorimetry and electrical bioimpedance, respectively. | 6 hours before SPECT acquisition.
  This study also aims to measure and compare the REE by indirect calorimetry with a Quark (Cosmed, Italy) calorimeter and the body composition by Byodinamics 450 (Biodynamics Corp., United States) within the two groups and across them.

CONTACTS AND LOCATIONS:
Overall Officials: Júlio S Marchini, Ph.D, Principal Investigator — Ribeirão Preto Medical School. São Paulo University (USP)
Locations (1):
- Clinical Hospital of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Goldstone AP. The hypothalamus, hormones, and hunger: alterations in human obesity and illness. Prog Brain Res. 2006;153:57-73. doi: 10.1016/S0079-6123(06)53003-1. PMID 16876568
- [Background] Figlewicz DP, Benoit SC. Insulin, leptin, and food reward: update 2008. Am J Physiol Regul Integr Comp Physiol. 2009 Jan;296(1):R9-R19. doi: 10.1152/ajpregu.90725.2008. Epub 2008 Oct 22. PMID 18945945
- [Background] Kishi T, Elmquist JK. Body weight is regulated by the brain: a link between feeding and emotion. Mol Psychiatry. 2005 Feb;10(2):132-46. doi: 10.1038/sj.mp.4001638. PMID 15630408
- [Background] Yun JW, Cho YK, Park JH, Kim HJ, Park DI, Sohn CI, Jeon WK, Kim BI. Abnormal glucose tolerance in young male patients with nonalcoholic fatty liver disease. Liver Int. 2009 Apr;29(4):525-9. doi: 10.1111/j.1478-3231.2008.01920.x. PMID 19323780
- [Background] Tataranni PA, DelParigi A. Functional neuroimaging: a new generation of human brain studies in obesity research. Obes Rev. 2003 Nov;4(4):229-38. doi: 10.1046/j.1467-789x.2003.00111.x. PMID 14649373
- [Background] DelParigi A, Chen K, Salbe AD, Reiman EM, Tataranni PA. Sensory experience of food and obesity: a positron emission tomography study of the brain regions affected by tasting a liquid meal after a prolonged fast. Neuroimage. 2005 Jan 15;24(2):436-43. doi: 10.1016/j.neuroimage.2004.08.035. PMID 15627585
- [Background] Matsuda M, Liu Y, Mahankali S, Pu Y, Mahankali A, Wang J, DeFronzo RA, Fox PT, Gao JH. Altered hypothalamic function in response to glucose ingestion in obese humans. Diabetes. 1999 Sep;48(9):1801-6. doi: 10.2337/diabetes.48.9.1801. PMID 10480611
- [Background] Suen VM, Silva GA, Tannus AF, Unamuno MR, Marchini JS. Effect of hypocaloric meals with different macronutrient compositions on energy metabolism and lung function in obese women. Nutrition. 2003 Sep;19(9):703-7. doi: 10.1016/s0899-9007(03)00104-7. PMID 12921877
- [Background] Nonino-Borges CB, Martins Borges R, Bavaresco M, Suen VM, Moreira AC, Marchini JS. Influence of meal time on salivary circadian cortisol rhythms and weight loss in obese women. Nutrition. 2007 May;23(5):385-91. doi: 10.1016/j.nut.2007.02.007. PMID 17483007
- [Background] Wichert-Ana L, Velasco TR, Terra-Bustamante VC, Araujo D Jr, Junior VA, Kato M, Leite JP, Assirati JA, MacHado HR, Bastos AC, Sakamoto AC. Typical and atypical perfusion patterns in periictal SPECT of patients with unilateral temporal lobe epilepsy. Epilepsia. 2001 May;42(5):660-6. doi: 10.1046/j.1528-1157.2001.41900.x. PMID 11380575
- See also: Record in the National Committee of Ethics in Research — http://portal2.saude.gov.br/sisnep/extrato_projeto.cfm?codigo=369688